CLINICAL TRIAL: NCT03882138
Title: Clinical Evaluation of Influence of Gingival Biotype on the Outcome of Open Flap Debridement in Patients With Chronic Periodontitis- An Interventional Study
Brief Title: Influence of Gingival Biotype on the Outcome of Open Flap Debridement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: perio bhumika
Record Dates: First submitted 2019-03-12; First posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thin biotype (Active Comparator): Modified Widman flap surgery followed by meticulous debridement, root planning and thorough irrigation with normal sterile saline solution
  Interventions: Procedure: open flap debridement
- thick biotype (Active Comparator): Modified Widman flap surgery followed by meticulous debridement, root planning and thorough irrigation with normal sterile saline solution
  Interventions: Procedure: open flap debridement

INTERVENTIONS:
Procedure: open flap debridement — Modified Widman flap surgery followed by meticulous debridement, root planning and thorough irrigation with normal sterile saline solution

SUMMARY:
The influence of periodontal thickness has been documented in outcome of various periodontal interventions like non surgical periodontal therapy, mucogingival therapy, guided tissue regeneration (GTR), crown lengthening and implant dentistry. There is lack of study showing the influence of gingival biotype on outcome of surgical procedure. The present study is therefore undertaken to evaluate the influence of gingival biotype on the outcome of open flap debridement for treatment of chronic periodontitis.

DETAILED DESCRIPTION:
Periodontitis is inflammation of the periodontal tissues resulting in clinical attachment loss, alveolar bone loss, and periodontal pocketing. Chronic periodontal disease can be successfully treated by non-surgical or surgical mechanical therapy provided adequate plaque control is maintained during the supportive phase of treatment. Elimination of these pockets by the therapist is necessary to allow the patient better access for plaque control. The goal of periodontal therapy, therefore, should include the creation of an oral environment in which the patient can cleanse every surface of every tooth. Ideally, this would be best accomplished by complete regeneration of the lost attachment apparatus and reestablishment of a minimal depth of sulcus.

It is seen that in pockets with shallow probing depths(1-3mm), there is reduction of pocket depth and loss of attachment by all the treatment modalities and more following surgical treatment. Lindhe et al. (1982) defined a critical probing depth below which the nonsurgical therapy is most likely to lead to loss of probing attachment In sites with moderate probing depth (4-6mm), there is more pocket reduction following MWF than subgingival curettage and SRP. Attachment gain is seen following all techniques and more following modified widman flap (MWF).

Deep pockets(>7mm) have shown reduction in probing depth following all the treatment modalities but more reduction is seen following MWF. More gain in attachment is seen following MWF than subgingival curettage.

Ramfjord observed an increase in pocket depth following periodontal treatment in shallow pockets. He also found loss of attachment with surgical therapy in moderate probing depth.

Histological findings in humans have revealed that there is loss of crestal bone as a consequence of periodontal surgical treatment. The resorption pattern varied with thickness of connective tissue covering the bone and was modified by injury to bone due to contact or near contact during instrumentation. Measurement indicated resorption occurs if retained tissue is 0.45 mm or less.

The influence of periodontal thickness has been documented in outcome of various periodontal interventions like non surgical periodontal therapy, mucogingival therapy, GTR, crown lengthening and implant dentistry.

Studies have shown that sites with thin gingiva lost attachment while no attachment loss is seen in sites with thick gingiva following non surgical therapy. Gingival thickness ≥0.8mm is associated with better root coverage with coronally advanced flap. Less recession is seen after GTR in sites with gingival thickness >1mm than the sites with <1mm. Thick biotype is also correlated with greater tissue rebound following surgical crown lengthening. Greater tissue recession is seen around implant with thin biotype.

Predictability of outcome following surgical procedures is of fundamental importance. Perusal of the available literature hints towards the need to further explore factors influencing the outcome of surgical procedures for the management of periodontitis. Periodontal biotype is one among such important factors.

The present study is therefore undertaken to evaluate the influence of gingival biotype on the outcome of open flap debridement for treatment of chronic periodontitis.

MATERIAL AND METHOD This study will be conducted in Department of Periodontics and Oral Implantology, Post Graduate Institute of Dental Sciences(PGIDS), Rohtak.

STUDY POPULATION Patients will be screened from outpatient department of Periodontics and Oral Implantology. The study will be conducted in 36 chronic periodontitis patients who had undergone phase 1 periodontal therapy.

Gingival biotype will be assessed by visibility of the periodontal probe through the gingival margin.

Group 1: Patient with thin biotype (periodontal probe is visible) Group 2: Patient with thick biotype (periodontal probe is not visible)

METHODOLOGY Periodontal examination Parameters recorded at baseline (on the day of surgery), at 3 months and 6 months follow up visit will be Plaque index (Silness and Loe) (PI) ; Gingival index (Loe and Silness) (GI); Bleeding on probing (BOP); Probing pocket depth (PPD); Clinical attachment level (CAL) and Gingival recession (REC). Probing pocket depth (PPD), Clinical attachment level (CAL). BOP will be assessed as a dichotomous measure (bleeding present or absent) within 15 seconds of probing. PPD will be recorded from gingival margin to base of pocket, and CAL from cementoenamel junction (CEJ) to base of pocket with university of North Carolina (UNC) 15 probe.

Methodology Patients meeting eligibility criteria will receive phase1 periodontal therapy consisting of scaling and root planing (SRP). SRP will be completed with ultrasonic scaler (EMS Piezon 250 ,Switzerland), hand scaler and curettes (Hu-Friedy) within two visits.

PERIODONTAL SURGICAL PROCEDURE After healing period of 8 weeks, clinical evaluation will be repeated and patients presenting atleast 4 residual periodontal pockets measuring ≥4 mm in maxillary or mandibular anterior segment will be subjected to surgical intervention. The study procedure will be explained to the patient in their own language. Written informed consent will be obtained from each patient.

Modified Widman flap surgery will be performed in both groups as described by Ramfjord and Nissle.37,38 After meticulous debridement, root planning and thorough irrigation with normal sterile saline solution, mucoperiosteal flaps will be repositioned and secured by using 3-0 black silk suture. Post operative instructions will be given.

POST OPERATIVE CARE Patients will be given both verbal and written instructions about post operative care including mouthrinse with 0.12% chlorhexidine digluconate solution twice daily for two weeks. All patient will be prescribed Amoxycillin 500mg thrice daily for 5 days and Ibuprofen 400 mg thrice daily for two days. Sutures will be removed after 1 week.

STATISTICAL ANALYSIS A minimum sample size of 18 patients in each group was calculated to be sufficient to detect a clinically important difference of 1mm gain in clinical attachment level with standard deviation of 1mm, 80% power of study and alpha level=0.05.To compensate for the expected dropouts in patient pool overtime, 20 patients will be involved in each group of this study.

Data recorded will be processed by standard statistical analysis. All statistical analysis will be carried out using statistical software (SPSS, Version 25.0 for Windows, SPSS, Chicago, IL).The normality of distribution of the data will be assessed using the Shapiro-Wilk test. . If it is in normal distribution, intra group comparison will be done by paired T test between two time points and inter group comparison will be done by using Independent T test between two groups. If it is in non normal distribution, intra group comparison will be done by Wilcoxon signed rank test and inter group comparison will be done by Mann-Whitney U test.. Statistical analysis of BOP will be done by McNemar test in intragroup and Chi-square test for intergroup comparison. Correlation and association between predictors and dependent variables will be analyzed by correlation analysis and regression analysis. Statistical significance level will be set at P≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients with moderate to severe chronic periodontitis
* Age 25-55 years
* Clinical attachment loss(CAL) ≥3 mm
* Probing pocket depth (PPD) ≥5 mm
* Possessing ≥20 natural teeth.

Exclusion Criteria:

* Patients with vertical bone loss
* Current or former smokers or use of tobacco in any form
* Pregnant women, lactating mothers and women taking oral contraceptives
* Patient who had undergone periodontal treatment within 6 months prior to the study
* Patient on anti-inflammatory drugs or antibiotics or history of treatment with medication known to influence periodontal status or healing such as statins, glucocorticoids, phenytoin, calcium channel blockers, immunosuppressants, bisphosphonates or any other host modulatory drug within six months of commencement of study
* Patient with average plaque index ≥1.5 after phase 1 therapy
* Miller Grade II /Grade III tooth mobility after SRP
* Periapical infection in any tooth of the surgical treatment segment.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
clinical attachment level | 6 months
  clinical attachment level is measured from cementoenamel junction to base of pocket

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No